CLINICAL TRIAL: NCT03663504
Title: A Randomised Study Comparing No Mechanical Bowel Preparation With Oral Antibiotics Alone in Patients Undergoing Elective Colon Surgery (REaCT-NSQIP)
Brief Title: Comparing No Mechanical Bowel Preparation With Oral Antibiotics Alone in Patients Undergoing Elective Colon Surgery
Acronym: REaCT-NSQIP
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OTT 18-03; REaCT-NSQIP (Other: Ottawa Hospital Research Institute)
Record Dates: First submitted 2018-08-07; First posted 2018-09-10 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Elective Colon Surgery
Keywords: Oral Antibiotics; Preoperative Mechanical Bowel Preparation; Surgical Site Infection; C. difficile
MeSH Terms: conditions — Surgical Wound Infection | interventions — preparation No. 012074; Neomycin; Metronidazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No Preparation (Active Comparator): No preparation before surgery
  Interventions: Other: No Preparation
- Oral Antibiotics (Active Comparator): Oral antibiotics (neomycin and flagyl), to be taken the day before the surgery
  Interventions: Drug: Neomycin and Flagyl

INTERVENTIONS:
Other: No Preparation — No preparation before surgery
  Arms: No Preparation
Drug: Neomycin and Flagyl — Oral antibiotic (Neomycin and Flagyl) taken the day before the surgery
  Other Names: Metronidazole
  Arms: Oral Antibiotics

SUMMARY:
The REaCT NSQIP will compare oral antibiotics vs. no antibiotics, which are two standards of care treatments for preoperative preparation of the bowel prior to colorectal surgery

DETAILED DESCRIPTION:
The divergence of clinical practice guidelines, in addition to observation from the large North American retrospective studies, suggest that surgeons and centers have not established a standard of care for the preoperative preparation of the bowel prior to colorectal surgery. Specifically, some centers are employing no preparation, others are administering a mechanical bowel preparation (MBP) and oral antibiotics and still others are using oral antibiotics alone. Recently, the Canadian Society of Colorectal Surgeons was unable to come to a consensus when attempting to update their preoperative guidelines because of the lack of agreement on best practice (personal communication). This is an important yet controversial topic in colorectal surgery and a clinical trial comparing two standard of care therapies will impact current practice in Canada. The REaCT-NSQIP study compares post-operative surgical infectious complications, length of stay, incidence of C. difficile rates, patient quality of life and cost-effectiveness in patients undergoing elective colorectal surgery with either no preparation or oral antibiotics. Data will be collected from the National Surgical Quality Improvement Program (NSQIP) and from patient quality of life questionnaires preoperatively and 30 days postoperatively

In this study, it is hypothesized that it is the oral antibiotics, and not the MBP, that is responsible for the reduction in postoperative infectious surgical complications (deep or superficial surgical site infection (SSI)) in patients undergoing elective colorectal resections. This improvement in postoperative infectious complications is not anticipated to result in a clinically significant increase in postoperative C. difficile infections or antibiotic resistant hospital-acquired infections.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective, non-emergency colon, resection surgery or abdominal perineal resection and no other requirements exists for a mechanical bowel preparation (as determined by the operating surgeon)
* 18 years of age or older
* Able to provide oral consent

Exclusion Criteria:

* Contraindication to the oral antibiotics, including allergies or adverse reactions to either metronidazole or neomycin
* Undergoing a rectal resection with a planned anastomosis (these patients will all receive MBP)
* Emergency surgery where no opportunity to administer preoperative oral antibiotics exists
* Requirement for a MBP (i.e. rectal resection with pelvic anastomosis, intraoperative colonoscopy, or at the discretion of the treating surgeon

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 630 (Actual)
Dates: Start 2018-10-23 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Post-Operative Surgical Infection Complication | 30 days
  To evaluate that use of oral antibiotics (neomycin and flagyl), administered the day prior to elective colonic resection is associated with a significant reduction in postoperative (within 30 days) surgical infectious complications (superficial and deep space infections).

SECONDARY OUTCOMES:
Grade III-IV Postoperative Surgical Site Infectious Complication | 30 days
  To evaluate the effects of oral antibiotics on Grade III-IV (Clavien-Dindo classification) postoperative surgical site infectious complication (at 30 days).
Postoperative Infections Complications | 30 days
  To evaluate the effects of oral antibiotics on postoperative infections complications classified as deep SSI, superficial SSI or non-SSI infectious complications (i.e. urinary tract infection, pneumonia, at 30 days).
Overall Postoperative Complication Rate | 30 days
  To evaluate the effects of oral antibiotics on overall postoperative complication rate (at 30 days).
Postoperative Length of Stay | Number of days spent in hospital post-operatively, average of 6 days
  To evaluate the effects of oral antibiotics on postoperative length of stay (LOS).
Incidence of Postoperative C. difficile Infections | 90 days
  To evaluate the effects of oral antibiotics on the incidence of postoperative C. difficile infections (at 90 days).
Incidence of Antibiotics Resistant Postoperative Infectious Complications | 30 days
  To evaluate the effects of oral antibiotics on the incidence of of antibiotics resistant postoperative infectious complications (at 30 days)
Patient Quality of Life | 30 days
  To evaluate the effects of oral antibiotics on patient quality of life by administering the SF-36 questionnaire, undertaken preoperatively and at 30 days postoperatively. The Short Form-36 (SF-36) is a 36-item, patient reported survey that is a measure of health status and commonly used in health economics. This SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. A low score denounces a worse outcome compared to a higher score that denounces a better outcome. The eight sections are: vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, emotional role functioning, social role functioning and mental health.
Direct Estimation of Health Utility Values | 30 days
  To evaluate the effects of oral antibiotics on patient quality of life by administering the EQ-5D-5L questionnaire, undertaken preoperatively and 30 days postoperatively. The EuroQol 5 Dimension 5 Level (EQ-5D-5L) questionnaire consists of two sections; the EQ-5D-5L descriptive system and the EQ Visual Analogue scale. The descriptive system comprises 5 dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression). There are 5 levels associated with it; no problems, slight problems, moderate problems, severe problems and extreme problems. The scale range of 1-5 is used for the 5 dimensions in the descriptive system where 1 is the best outcome and 5 is the worst outcome. The Visual Analogue scale records the respondent's self-rated health on a vertical, visual scale with endpoints labelled 'the best health you can imagine' at the top and 'the worst health you can imagine' at the bottom. This ranges 0 being the worst outcome to 100 being the best outcome.
Incremental Cost-Effectiveness Ratio | Through to study completion, an average of 2 years
  To evaluate the effects of antibiotics on the incremental cost-effectiveness ratio

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Auer, MD, Principal Investigator — Ottawa Hospital Research Institute; Sameer Apte, MD, Principal Investigator — The Ottawa Hospital
Locations (6):
- Canada (6):
  - The Queen Elizabeth II Health Sciences Centre, Halifax, Nova Scotia
  - The Ottawa Hospital Cancer Centre, Ottawa, Ontario
  - Hôpital Montfort, Ottawa, Ontario
  - Queensway Carleton Hospital, Ottawa, Ontario
  - Renfrew Victoria Hospital, Renfrew, Ontario
  - University Health Network, Toronto, Ontario

REFERENCES:
- [Background] Apte SS, Moloo H, Jeong A, Liu M, Vandemeer L, Suh K, Thavorn K, Fergusson DA, Clemons M, Auer RC. Prospective randomised controlled trial using the REthinking Clinical Trials (REaCT) platform and National Surgical Quality Improvement Program (NSQIP) to compare no preparation versus preoperative oral antibiotics alone for surgical site infection rates in elective colon surgery: a protocol. BMJ Open. 2020 Jul 9;10(7):e036866. doi: 10.1136/bmjopen-2020-036866. PMID 32647023
- [Derived] Willis MA, Toews I, Soltau SL, Kalff JC, Meerpohl JJ, Vilz TO. Preoperative combined mechanical and oral antibiotic bowel preparation for preventing complications in elective colorectal surgery. Cochrane Database Syst Rev. 2023 Feb 7;2(2):CD014909. doi: 10.1002/14651858.CD014909.pub2. PMID 36748942
- See also: The Rethinking Clinical Trials (REaCT) website — https://react.ohri.ca/